CLINICAL TRIAL: NCT03077256
Title: Multicenter Prospective Registry to Evaluate Use and Outcomes of Burst Biologics Products in Foot and Ankle Surgery
Brief Title: Burst Biologics Foot and Ankle Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Burst Biologics (Industry)
Responsible Party: Sponsor-Investigator, Burst Biologics, Medical Affairs Officer, Smart-Surgical Inc. dba Burst Biologics
Organization: Smart-Surgical Inc. dba Burst Biologics (Industry)
Other Study IDs: FA002
Record Dates: First submitted 2017-02-13; First posted 2017-03-10 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Foot and Ankle Disorders; Ankle Fusion, Osteotomy
Keywords: Ankle Arthrodesis; Cellular Allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BioBurst Fluid, Burst Allograft — BioBurst Fluid, Burst Allograft in Foot and Ankle Surgery

SUMMARY:
This prospective registry was designed as an observational study to ascertain how commercially available Burst Products are being used by foot and ankle surgeons performing procedures which involve bone grafting, as well as determining relevant patient outcomes.

DETAILED DESCRIPTION:
Foot and ankle surgery requiring the use of bone graft is common despite recent advancements and improved outcomes with new motion preservation devices (ankle replacement). Autogenous bone remains the gold standard but is complicated by donor site morbidity and availability of a sufficient volume of graft. Over the past two decades surgeon interest in alternative bone grafts has steadily increased. Bone morphogenic proteins, synthetic bone graft substitutes, and various allograft products are widely available to surgeons. Limitations on the use of allografts in the past were mainly attributed to less than optimal donor screening and processing techniques which removed viable components needed to aid in the bone healing process.

In recent years, the focus and scientific advances in various allograft processing techniques have allowed the retention of various viable cytokines, growth factors, and cell populations which result in enhanced osteogenic and osteoinductive properties. Rigorous donor bone screening and meticulous testing has virtually eliminated the risk of disease transmission.

A unique proprietary cryoprotection processing technique for allograft tissue was developed by Smart-Surgical, Inc. and a complete line of allograft products was created and is now marketed by Burst Biologics (dba). In addition, rigorous standardized laboratory assay techniques and statistical analysis provide consistency and uniformity of the biologically active components of Burst allograft products.

This prospective registry was designed as an observational study to ascertain how commercially available Burst Products are being used by foot and ankle surgeons performing procedures which involve bone grafting, as well as determining relevant patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient diagnosed with a pathology of the hindfoot, foot, or ankle requiring surgical intervention.
* The surgeon has determined that a Burst Biologic product is or was clinically indicated.
* Patient capable of understanding the content of the Informed Consent Form.
* Patient willing and able to participate in the registry protocol including the surgeon's standard follow-up visits and clinical evaluations.
* Patient who has agreed to participate in the registry by providing consent per the applicable local law and the declaration of Helsinki.

Exclusion Criteria: The following are relative contraindications for the use of Burst Products, however the investigator surgeon is solely responsible for the determination of patient eligibility for surgery:

* Severe vascular or neurological disease
* Uncontrolled diabetes
* Severe degenerative disease (other than degenerative disc disease)
* Hypercalcemia, abnormal calcium metabolism
* Existing acute or chronic infections, especially at the site of the operation
* Inflammatory bone disease such as osteomyelitis
* Malignant tumors
* Patients who are or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the study will be drawn from the individual surgeons practice. Patients will be either candidates for foot and ankle surgery after having failed conservative treatment or will have had foot and ankle surgery and the surgeon determined that the use of a Burst Biologic product is or was clinically indicated. Only patients who consent to participate and meet the inclusion-exclusion criteria will be included provided that a Burst Biologic product will be used in the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Fusion (%) Number of fusion patients fused/all fusion patients operated | 6 Months
  Determined by CT Scan or Plain Radiographs
Bone Consolidation (%) Number of osteotomy patients with bone consolidation/all osteotomy patients operated | 6 Months
  Determined by CT Scan or Plain Radiographs

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 6 Months
Change from Baseline in American Orthopedic Foot and Ankle Society Questionnaire (AOFAS) Score | 6 Months
Change from Baseline in Foot Function Index Score (FFI) | 6 Months
Change from Baseline in Short Form-36 V2 | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Czop, R.Ph., Study Director — Medical Affairs Officer
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No